CLINICAL TRIAL: NCT03823898
Title: Lifestyle Intervention in Overweight and Obese Premenopausal Women
Brief Title: Lifestyle Intervention in Overweight Women
Acronym: PESO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Motricidade Humana (Other)
Responsible Party: Principal Investigator, Luís Bettencourt Sardinha, Principal investigator, Faculdade de Motricidade Humana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PESO-2002
Record Dates: First submitted 2019-01-27; First posted 2019-01-31 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Weight Loss; Lifestyle, Sedentary; Physical Activity; Nutritional and Metabolic Disease; Behavior, Health; Cardiovascular Risk Factor
Keywords: obesity; body composition; weight management; cardiovascular and metabolic markers; Behavioral change; Exercise
MeSH Terms: conditions — Obesity; Weight Loss; Sedentary Behavior; Motor Activity; Metabolic Diseases; Health Behavior

STUDY DESIGN:
Intervention Model Description: A clinical trial with three-arm
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised exercise (Experimental): Participants in this group received a lifestyle intervention from baseline to 4 months. From 4 to 16 months participants were involved in two supervised exercise sessions per week plus healthy lifestyle interactive sessions.
  The experimental intervention consisted of: a) monthly behavioral sessions consisted of lifestyle interactive sessions took place monthly and covered and followed contents that were addressed during the first 4 months of the study; b) The supervised exercise sessions were prescribed using an aerobic mode performed at a moderate-to-vigorous intensity during 45 minutes, twice a week, preferably during the weekends.
  Interventions: Behavioral: Supervised exercise; Behavioral: Lifestyle intervention from baseline to 4 months; Behavioral: Monthly behavioral sessions
- Control Group (Active Comparator): Participants in this group received a lifestyle intervention from baseline to 4 months. From 4 to 16 months participants received no intervention
  Interventions: Behavioral: Lifestyle intervention from baseline to 4 months
- Monthly behavioral sessions (Experimental): Participants in this group received a lifestyle intervention from baseline to 4 months and then from 4 to 16 months participants were involved in non-supervised exercise group sessions with monthly behavioral sessions.
  The experimental intervention consisted of monthly behavioral sessions consisted of lifestyle interactive sessions took place monthly and covered and followed contents that were addressed during the first 4 months of the study
  Interventions: Behavioral: Lifestyle intervention from baseline to 4 months; Behavioral: Monthly behavioral sessions

INTERVENTIONS:
Behavioral: Supervised exercise — Two supervised exercise sessions per week from months 4 to 16
  Arms: Supervised exercise
Behavioral: Lifestyle intervention from baseline to 4 months — Lifestyle intervention from baseline to 4 months
Behavioral: Monthly behavioral sessions — Monthly behavioral sessions consisted of lifestyle interactive sessions will take place monthly and covered and followed contents that were addressed during the first 4 months of the study
  Arms: Monthly behavioral sessions; Supervised exercise

SUMMARY:
The Exercise and Obesity Health Promotion (PESO) program is a randomized controlled trial designed to analyze the effects of a lifestyle intervention in weight management and health-related parameters of overweight and obese premenopausal women

DETAILED DESCRIPTION:
The PESO (Exercise and Obesity Health Promotion Program) is a program of weight control and exercise promotion for overweight and obese premenopausal women, developed by specialists in exercise, nutrition, and psychology, under medical supervision. It is a program that promotes the autonomy of the participants and the permanent modification of their habits and lifestyles, without the use of drugs or any other products, devices, or techniques of "slimming".

Participants in the PESO Program were able to enjoy a regular and multifaceted group program, aiming to increase knowledge about permanent body weight control, increased motivation and practice of physical activity and exercise, and improved habits food and nutrition. Increases in functional mobility, metabolic health, quality of life and the physical and mental well-being of the participants are central priorities of this Program.

The PESO Program was conducted in a university context and was led by teachers and researchers from the Faculty of Human Motors and other national and foreign institutions. The program is not for commercial purposes, it does not entail financial costs for the participants and it is involved in a wide range of scientific research projects, which have been recognized by individuals and external entities as relevant and of interest to the general population and the community in particular.

ELIGIBILITY:
Inclusion Criteria:

* older than 24 years,
* be premenopausal and not currently pregnant,
* BMI higher than 24.9 kg/m2,
* free from major disease

Exclusion Criteria:

* Not meeting the inclusion criteria

Ages: 24 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2002-01-02 (Actual); Primary Completion 2003-07-01 (Actual); Study Completion 2003-12-01 (Actual)

PRIMARY OUTCOMES:
Body weight | 0 months
  A scale (Seca, Hamburg, Germany) was used to assess body weight
Body weight | 4 months
  A scale (Seca, Hamburg, Germany) was used to assess body weight
Body weight | 16 months
  A scale (Seca, Hamburg, Germany) was used to assess body weight
Body weight | 22 months
  A scale (Seca, Hamburg, Germany) was used to assess body weight

SECONDARY OUTCOMES:
Body height | 0 months
  A scale (Seca, Hamburg, Germany) was used to determine body height
total and regional fat and fat-free mass | 0 months
  Dual-energy x-ray absorptiometry (pencil beam mode, QDR-1500 Hologic, United States) was used to assess changes in total and regional fat and fat-free mass.
total and regional fat and fat-free mass | 4 months
  Dual-energy x-ray absorptiometry (pencil beam mode, QDR-1500 Hologic, United States) was used to assess changes in total and regional fat and fat-free mass.
total and regional fat and fat-free mass | 16 months
  Dual-energy x-ray absorptiometry (pencil beam mode, QDR-1500 Hologic, United States) was used to assess changes in total and regional fat and fat-free mass.
Thigh Adipose Tissue | 0 months
  Using the same scan parameters, contiguous 7-mm-thick cross-sectional images of both legs were obtained between the inferior ischial tuberosity and the superior border of the patella. Total/subcutaneous thigh Adipose tissue was measured by axial computerized tomography (Somaton Plus; Siemens, Germany).
Thigh Adipose Tissue | 16 months
  Using the same scan parameters, contiguous 7-mm-thick cross-sectional images of both legs were obtained between the inferior ischial tuberosity and the superior border of the patella. Total/subcutaneous thigh Adipose tissue was measured by axial computerized tomography (Somaton Plus; Siemens, Germany).
Thigh Muscle Distribution | 0 months
  Using the same scan parameters, contiguous 7-mm-thick cross-sectional images of both legs were obtained between the inferior ischial tuberosity and the superior border of the patella. Muscle tissue was measured by axial computerized tomography (Somaton Plus; Siemens, Germany).
Thigh Muscle Distribution | 16 months
  Using the same scan parameters, contiguous 7-mm-thick cross-sectional images of both legs were obtained between the inferior ischial tuberosity and the superior border of the patella. Muscle tissue was measured by axial computerized tomography (Somaton Plus; Siemens, Germany).
Abdominal Adipose Tissue Distribution | 0 months
  With the subjects supine and arms extended above their head, a single cross-sectional axial computerized tomography (Somaton Plus; Siemens, Germany) L4-L5 intervertebral space image was acquired to measure abdominal adipose tissue compartments
Abdominal Adipose Tissue Distribution Changes | 16 months
  With the subjects supine and arms extended above their head, a single cross-sectional axial computerized tomography (Somaton Plus; Siemens, Germany) L4-L5 intervertebral space image was acquired to measure abdominal adipose tissue compartments
triglycerides | 0 months
  An enzymatic colorimetric method was used to determine triglycerides
triglycerides | 16 months
  An enzymatic colorimetric method was used to determine triglycerides
uric acid | 0 months
  An enzymatic colorimetric method was used to determine uric acid
uric acid | 16 months
  An enzymatic colorimetric method was used to determine uric acid
total cholesterol | 0 months
  An enzymatic colorimetric method was used to determine total cholesterol
total cholesterol | 16 months
  An enzymatic colorimetric method was used to determine total cholesterol
low-density lipoprotein cholesterol | 0 months
  An enzymatic colorimetric method was were used to determine low-density lipoprotein cholesterol
low-density lipoprotein cholesterol | 16 months
  An enzymatic colorimetric method was were used to determine low-density lipoprotein cholesterol
high-density lipoprotein cholesterol | 0 months
  An enzymatic colorimetric method was used to determine high-density lipoprotein cholesterol
high-density lipoprotein cholesterol | 16 months
  An enzymatic colorimetric method was used to determine high-density lipoprotein cholesterol
Cardiorespiratory | 0 months
  A graded exercise testing with gases analysis was used to assess cardio-respiratory changes
Cardio-respiratory | 16 months
  A graded exercise testing with gases analysis was used to assess cardio-respiratory changes
Total-body water | 0 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess total-body water
Total-body water | 16 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess total-body water
Extracellular water | 0 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess extracellular water
Extracellular water | 16 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess extracellular water
Intracellular water | 0 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess intracellular water
Intracellular water | 16 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess intracellular water
Resistance | 0 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess resistance
Resistance | 16 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess resistance
Reactance | 0 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess reactance
Reactance | 16 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess reactance
Phase angle | 0 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess phase angle
Phase angle | 16 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess phase angle
Bioelectrical Impedance Vector Analysis | 0 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess changes in Bioelectrical Impedance Vector Analysis
Bioelectrical Impedance Vector Analysis | 16 months
  Bioelectrical impedance spectroscopy (Hydra 4200 Xitron, United States) was used to assess changes in Bioelectrical Impedance Vector Analysis
Quality of life reported | 0 months
  The quality of life was reported through the SF-36 questionnaire. The SF-36 is a 36-item, generic quality-of-life measure that assesses 8 domains: (1) physical functioning; (2) role limitation due to physical-health problems; (3) bodily pain; (4) general health perceptions; (5) vitality; (6) social functioning; (7) role limitations due to emotional-health problems; and (8) mental health. Social function, vitality, and general health perceptions scales measure both physical and mental health status. All health measures were scored on scales of 0 to 100, with higher scores indicating better health.
Quality of life reported | 4 months
  The quality of life was reported through the SF-36 questionnaire. The SF-36 is a 36-item, generic quality-of-life measure that assesses 8 domains: (1) physical functioning; (2) role limitation due to physical-health problems; (3) bodily pain; (4) general health perceptions; (5) vitality; (6) social functioning; (7) role limitations due to emotional-health problems; and (8) mental health. Social function, vitality, and general health perceptions scales measure both physical and mental health status. All health measures were scored on scales of 0 to 100, with higher scores indicating better health.
Quality of life reported | 16 months
  The quality of life was reported through the SF-36 questionnaire. The SF-36 is a 36-item, generic quality-of-life measure that assesses 8 domains: (1) physical functioning; (2) role limitation due to physical-health problems; (3) bodily pain; (4) general health perceptions; (5) vitality; (6) social functioning; (7) role limitations due to emotional-health problems; and (8) mental health. Social function, vitality, and general health perceptions scales measure both physical and mental health status. All health measures were scored on scales of 0 to 100, with higher scores indicating better health.
Blood pressure | 0 months
  A sphygmomanometer was used to determine changes in systolic and diastolic blood pressure
Blood pressure | 16 months
  A sphygmomanometer was used to determine changes in systolic and diastolic blood pressure
Physical activity | 0 months
  A self-reported measure of physical activity was used, specifically the short-form of the International physical activity questionnaire (IPAQ-SF). The IPAQ-SF records the last 7 day recall for four intensity levels of physical activity which is vigorous-intensity activity, moderate-intensity activity, walking, and sitting. From IPAQ data were converted to Metabolic Equivalent minutes per week (MET-min/week) using the published formulation the Compendium average MET score. Physical activity of low intensity was characterized by activities inducing less than 3 metabolic equivalents (MET), moderate intensity between 3 and 5.9 MET and for vigorous intensity higher than 6 MET. The higher the number of MET, the higher the intensity. The duration of the activities in each intensity were calculated based on the reported time per week. The higher the duration in activities of moderate to vigorous physical activity the highest the physical activity level
Physical activity | 4 months
  A self-reported measure of physical activity was used, specifically the short-form of the International physical activity questionnaire (IPAQ-SF). The IPAQ-SF records the last 7 day recall for four intensity levels of physical activity which is vigorous-intensity activity, moderate-intensity activity, walking, and sitting. From IPAQ data were converted to Metabolic Equivalent minutes per week (MET-min/week) using the published formulation the Compendium average MET score. Physical activity of low intensity was characterized by activities inducing less than 3 metabolic equivalents (MET), moderate intensity between 3 and 5.9 MET and for vigorous intensity higher than 6 MET. The higher the number of MET, the higher the intensity. The duration of the activities in each intensity were calculated based on the reported time per week. The higher the duration in activities of moderate to vigorous physical activity the highest the physical activity level
Physical activity | 16 months
  A self-reported measure of physical activity was used, specifically the short-form of the International physical activity questionnaire (IPAQ-SF). The IPAQ-SF records the last 7 day recall for four intensity levels of physical activity which is vigorous-intensity activity, moderate-intensity activity, walking, and sitting. From IPAQ data were converted to Metabolic Equivalent minutes per week (MET-min/week) using the published formulation the Compendium average MET score. Physical activity of low intensity was characterized by activities inducing less than 3 metabolic equivalents (MET), moderate intensity between 3 and 5.9 MET and for vigorous intensity higher than 6 MET. The higher the number of MET, the higher the intensity. The duration of the activities in each intensity were calculated based on the reported time per week. The higher the duration in activities of moderate to vigorous physical activity the highest the physical activity level
Energy intake | 0 months
  Energy intake was assessed during a 3-day period by a 24-hour diet record. Subjects were instructed regarding portion sizes, supplements, food preparation aspects, and other aspects pertaining to an accurate recording of their energy intake. Records were turned in and reviewed at the time of laboratory testing for total energy intake. Dietary records were analyzed using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Energy intake | 4 months
  Energy intake was assessed during a 3-day period by a 24-hour diet record. Subjects were instructed regarding portion sizes, supplements, food preparation aspects, and other aspects pertaining to an accurate recording of their energy intake. Records were turned in and reviewed at the time of laboratory testing for total energy intake. Dietary records were analyzed using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Energy intake | 16 months
  Energy intake was assessed during a 3-day period by a 24-hour diet record. Subjects were instructed regarding portion sizes, supplements, food preparation aspects, and other aspects pertaining to an accurate recording of their energy intake. Records were turned in and reviewed at the time of laboratory testing for total energy intake. Dietary records were analyzed using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Macro-nutrient | 0 months
  Macro-nutrient intake was assessed during a 3-day period by a 24-hour diet record. Subjects were instructed regarding portion sizes, supplements, food preparation aspects, and other aspects pertaining to an accurate recording of their food intake. Records were turned in and reviewed at the time of laboratory testing. Dietary records were analyzed using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Macro-nutrient | 4 months
  Macro-nutrient intake was assessed during a 3-day period by a 24-hour diet record. Subjects were instructed regarding portion sizes, supplements, food preparation aspects, and other aspects pertaining to an accurate recording of their food intake. Records were turned in and reviewed at the time of laboratory testing. Dietary records were analyzed using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Macro-nutrient | 16 months
  Macro-nutrient intake was assessed during a 3-day period by a 24-hour diet record. Subjects were instructed regarding portion sizes, supplements, food preparation aspects, and other aspects pertaining to an accurate recording of their food intake. Records were turned in and reviewed at the time of laboratory testing. Dietary records were analyzed using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Micro-nutrient | 0 months
  Micronutrient intake was assessed during a 3-day period by a 24-hour diet record. Subjects were instructed regarding portion sizes, supplements, food preparation aspects, and other aspects pertaining to an accurate recording of their food intake. Records were turned in and reviewed at the time of laboratory testing. Dietary records were analyzed using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Micro-nutrient | 4 months
  Micronutrient intake was assessed during a 3-day period by a 24-hour diet record. Subjects were instructed regarding portion sizes, supplements, food preparation aspects, and other aspects pertaining to an accurate recording of their food intake. Records were turned in and reviewed at the time of laboratory testing. Dietary records were analyzed using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Micro-nutrient | 16 months
  Micronutrient intake was assessed during a 3-day period by a 24-hour diet record. Subjects were instructed regarding portion sizes, supplements, food preparation aspects, and other aspects pertaining to an accurate recording of their food intake. Records were turned in and reviewed at the time of laboratory testing. Dietary records were analyzed using a software package (Food Processor SQL, ESHA Research, Salem, OR, USA).
Resting Metabolic rate | 0 months
  Indirect calorimetry for determining resting metabolic rate
Resting Metabolic rate | 16 months
  Indirect calorimetry for determining resting metabolic rate
Anthropometric (circumferences) | 0 months
  An anthropometric tape was used to measure body circumferences
Anthropometric (circumferences) | 4 months
  An anthropometric tape was used to measure body circumferences
Anthropometric (circumferences) | 16 months
  An anthropometric tape was used to measure body circumferences
Anthropometric (skinfolds) | 0 months
  A caliper was used to measure skinfolds
Anthropometric (skinfolds) | 4 months
  A caliper was used to measure skinfolds
Anthropometric (skinfolds) | 16 months
  A caliper was used to measure skinfolds
Fasting insulin | 0 months
  Electrochemiluminescence immunoassay (ECLIA) was used to assess fasting insulin
Fasting insulin | 16 months
  Electrochemiluminescence immunoassay (ECLIA) was used to assess fasting insulin
Fasting glycemia | 0 months
  Fasting glycemia was assessed by hexokinase method
Fasting glycemia | 16 months
  Fasting glycemia was assessed by hexokinase method
Interleukin-6 | 0 months
  Interleukin-6 (IL-6) was measured by chemiluminescence immunoassay
Interleukin-6 | 16 months
  Interleukin-6 (IL-6) was measured by chemiluminescence immunoassay
Tumor necrosis factor-alpha | 0 months
  Tumor necrosis factor-alpha (TNF-alpha) was measured using a high-sensitivity enzyme linked immunosorbent assay (ELISA) principle
Tumor necrosis factor-alpha | 16 months
  Tumor necrosis factor-alpha (TNF-alpha) was measured using a high-sensitivity enzyme linked immunosorbent assay (ELISA) principle
Plasminogen activator inhibitor-1 | 0 months
  Plasminogen activator inhibitor-1 (PAI-1) was measured in iced citrated plasma using the Coatest PAI method (enzyme immunoassay-EIA)
Plasminogen activator inhibitor-1 | 16 months
  Plasminogen activator inhibitor-1 (PAI-1) was measured in iced citrated plasma using the Coatest PAI method (enzyme immunoassay-EIA)
fibrinogen concentrations | 0 months
  Fibrinogen concentrations were measured by clotting time
fibrinogen concentrations | 16 months
  Fibrinogen concentrations were measured by clotting time
Hemoglobin A1c | 0 months
  Hemoglobin A1c (Hb A1c) was determined by high-pressure liquid chromatography (HPLC)
Hemoglobin A1c | 16 months
  Hemoglobin A1c (Hb A1c) was determined by high-pressure liquid chromatography (HPLC)
serum adiponectin concentration | 0 months
  Serum adiponectin concentration was measured by radioimmunoassay (RIA)
serum adiponectin concentration | 16 months
  Serum adiponectin concentration was measured by radioimmunoassay (RIA)
serum leptin concentration | 0 months
  Serum leptin concentration was measured by radioimmunoassay (RIA)
serum leptin concentration | 16 months
  Serum leptin concentration was measured by radioimmunoassay (RIA)
urine cortisol | 0 months
  Urine cortisol was measured by radioimmunoassay (RIA)
urine cortisol | 16 months
  Urine cortisol was measured by radioimmunoassay (RIA)
microalbuminuria | 0 months
  Microalbuminuria plasma concentration was measured by high-sensitivity particle-enhanced turbidimetric assay
microalbuminuria | 16 months
  Microalbuminuria plasma concentration was measured by high-sensitivity particle-enhanced turbidimetric assay
C-reactive protein | 0 months
  C-reactive protein plasma concentration was measured by high-sensitivity particle-enhanced turbidimetric assay
C-reactive protein | 16 months
  C-reactive protein plasma concentration was measured by high-sensitivity particle-enhanced turbidimetric assay
apolipoprotein A1 | 0 months
  Apolipoprotein A1 plasma concentration was measured by high-sensitivity particle-enhanced turbidimetric assay
apolipoprotein A1 | 16 months
  Apolipoprotein A1 plasma concentration was measured by high-sensitivity particle-enhanced turbidimetric assay
apolipoprotein B100 | 0 months
  Apolipoprotein B100 plasma concentration was measured by high-sensitivity particle-enhanced turbidimetric assay
apolipoprotein B100 | 16 months
  Apolipoprotein B100 plasma concentration was measured by high-sensitivity particle-enhanced turbidimetric assay
Alanine aminotransferase | 0 months
  Alanine aminotransferase was determined by a kinetic method
Alanine aminotransferase | 16 months
  Alanine aminotransferase was determined by a kinetic method
Aspartate aminotransferase | 0 months
  Aspartate aminotransferase was determined by a kinetic method
Aspartate aminotransferase | 16 months
  Aspartate aminotransferase was determined by a kinetic method

CONTACTS AND LOCATIONS:
Overall Officials: Luís B Sardinha, PhD, Study Director — Faculdade Motricidade Humana
Locations (1):
- Faculdade de Motricidade Humana, Oeiras, Cruz-Quebrada, Portugal

IPD SHARING:
Plan to Share IPD: No
No plans for IPD